CLINICAL TRIAL: NCT00325585
Title: Couples HIV Intervention Randomized Controlled Trial
Brief Title: HIV Prevention Intervention for Couples
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01DA015641 (NIH); R01DA015641 (NIH)
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Human Immunodeficiency Viruses; Acquired Immunodeficiency Syndrome; Substance Abuse; Sexually Transmitted Disease, Viral; Intervention Studies; Women's Health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Sexually Transmitted Diseases, Viral

INTERVENTIONS:
Behavioral: Couples HIV counseling and testing
Behavioral: Women's relationship-focused HIV counseling and testing

SUMMARY:
Recent studies have shown that many drug-using minority women are vulnerable to HIV infection from their husbands or other intimate male partners. The goal of this study is to develop and evaluate two new HIV counseling and testing programs designed for drug-using women at risk for HIV from a primary male partner. It is predicted that HIV counseling and testing programs administered to couples rather than to women only, and programs that focus on intimate relationships in the context of HIV risk, will result in a reduction of risky sexual and drug-related behavior among drug-using women and their primary male partners. This four-year study employs a randomized clinical trial (RCT) design to test the effectiveness of two new HIV counseling and testing programs for women drug-users in Harlem and the South Bronx in New York City.

DETAILED DESCRIPTION:
The broad, long-term objective of this research is to establish primary preventive interventions to reduce human immunodeficiency virus (HIV) risk behavior among drug-using minority women. Recent studies indicate that high rates of sexual risk behavior occur within drug-using minority women's primary heterosexual relationships. Based on an integrated theory of HIV risk behavior, it is predicted that (a) interventions administered to couples rather than to women only, and (b) interventions that focus on relationship dynamics in the context of HIV risk, will result in a reduction of sexual and drug-related risk behavior among drug-using women and their primary partners. This four-year study employs a randomized clinical trial (RCT) 3-group design to test the efficacy of HIV intervention modality (couples versus women-only) and intervention content (relationship-focused versus standard HIV counseling and testing) on crack, cocaine and heroin (injected and noninjected) using women's sexual risk with primary partners.

A total of 390 women drug-users and their partners are recruited from the streets of Harlem and the South Bronx in New York City. Participants are randomly assigned to one of three HIV counseling and testing intervention conditions: (a) couples, relationship-focused; (b) women-only, relationship-focused; or, (c) NIDA women-only standard HIV-CT (control). All subjects are administered baseline, 3-month, and 9-month follow-up assessments using a combination of computer-assisted personal interview (CAPI) and computer-assisted self interview (CASI) techniques. In addition to sociodemographic characteristics, the interview will measure drug-use patterns, HIV risk behavior, and dyadic- and individual-level variables operationalized to test specific hypotheses of women's HIV risk behavior and behavior change. In addition to testing the effectiveness of the experimental interventions, data analyses will determine the theory-driven psychosocial mechanisms that act to mediate and moderate any observed association between intervention treatment and subsequent risk reduction. Incremental cost-effectiveness analyses will also be performed.

Results from this study will allow researchers to determine whether couple-based HIV counseling and testing is a more effective (and cost-effective) approach to HIV prevention than individual HIV counseling and testing. Analyses will further provide information on the specific components of couple-based interventions that were most effective in reducing HIV risk behavior, thereby contributing to theory development regarding intimate couples' HIV risk.

ELIGIBILITY:
Inclusion Criteria:

For women:

* 18 years of age or older
* self-reported use of crack, cocaine or heroin in prior 30 days
* has male sex partner identified as primary partner for at least one year
* had unprotected vaginal or anal sex with current partner in prior 30 days
* able to enlist partner in study enrollment
* would not feel threatened participating in the study with primary partner
* must not have participated in HIV/AIDS related study or attended HIV counseling and testing session in six months
* self-reported HIV negative or sero-unaware

For men:

* 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
risk behaviors

CONTACTS AND LOCATIONS:
Overall Officials: James M McMahon, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- NDRI South Bronx Field Office, The Bronx, New York, United States